CLINICAL TRIAL: NCT01469403
Title: Weight Loss Intervention Before Total Knee Replacement, a Randomized Controlled Trial
Brief Title: Weight Loss Intervention Before Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Rheumatism Association (Other); Cambridge Weight Plan Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TKABMI
Record Dates: First submitted 2011-09-07; First posted 2011-11-10 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2011-11

CONDITIONS: Osteoarthritis, Knee; Obesity
Keywords: Osteoarthritis, knee; Obesity; Weight Loss; Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Weight Loss | interventions — Weight Reduction Programs

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): Standard procedure for knee arthroplasty
- Weight loss program (Active Comparator): The intervention program consists of 8 weeks of low-diet, using formula foods, and dietary counseling before surgery. When using formula foods the patients can achieve a quicker weight reduction and a greater reduction in fat mass than using conventional dietetic hypo caloric diet.
  Interventions: Behavioral: 8 weeks weight loss program, Cambridge.

INTERVENTIONS:
Behavioral: 8 weeks weight loss program, Cambridge. — Fast weight losses improve the prognosis for the sustained weight loss. During the first week a dietitian will tutor the participants in formula food diet (The Cambridge Health and Weight plan UK.), followed by seven weeks with control guidance and instruction in healthy eating habits once a week. The guidance by the dietitian will be carried out both on an individual basis and in groups. The goal of the intervention is to achieve a preoperative weight loss of at least 5 to 10% of the patient's body weight, thus improving patient's health before surgery.
  Arms: Weight loss program

SUMMARY:
The purpose of this study is to compare the efficacy in a group of patients who must follow the current procedure for treatment of artificial knee, compared with a group of patients who must undergo an 8-week weight loss program before surgery. 1 year after surgery the investigators will examine whether there are differences between the two groups' quality of life and functional capacity.

DETAILED DESCRIPTION:
Background In Denmark the numbers of primary total knee arthroplasty (TKA) operations annually increase. In the year 2000 was performed approximately 2,500 operations and in 2008 was performed more than 7,500 total knee arthroplasty operations, and there appears in all countries to be similar tendency. Meanwhile, the prevalence of overweight and obesity has increased markedly over the last 50 years. Approximately 13% of the Danish population is obese. For several years the association between obesity and knee osteoarthritis (OA) has been recognized, and osteoarthritis is the most frequent indication for total knee arthroplasty(80%).

The purpose of this study is to investigate whether weight loss interventions before primary total knee arthroplasty will improve quality of life and functional level, reduce pain and risk of early and late postoperative complications.

Sample size Significance level is set to 5% by using a 2-sided analysis and the power is set at 80%. Based on an expectation of a difference in patient-reported outcome scores in between the groups at 8%, as measured by SF-36 12 months postoperatively, standard deviation (SD) 13 must be include 41 participants in each group. To allow a drop-out rate of 20% the group size increases to 51 participants in each group. In total 102 participants.

Statistical analysis, The two groups scores at 12 months postoperatively, and the two groups' change in the primary outcome measurer, from 1 week before surgery to 12 months postoperatively, compared with t-test or Mann-Whitney test rang sum depending on data distribution.

ELIGIBILITY:
Inclusion Criteria:

* All patients recommended for primary total knee replacement.
* Body mass index > 30.
* Must be motivated for weight loss.
* Must be able to read and understand Danish.

Exclusion Criteria:

* Rheumatoid arthritis.
* Patients who are operated on both knees during the project period can only participate once.
* Planned obesity surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
SF-36 | Measured 12 months postoperatively.
  A patient reported outcome (PRO). The questionnaire is a tool for measuring health status. The form is used to measure the patient's view of his own health by scoring standardized responses to standardized questions. The schedule consists of 36 questions representing eight health concepts.

SECONDARY OUTCOMES:
6 minutes walk test (6MW). | Measured 1 week before surgery.
  Used to target the operating level of the patient's daily activities.
Body composition | Measured 1 week before surgery.
  Dual energy X-ray absorptiometry (DEXA) can measure total body bone mineral density and obtain accurate measurements of body tissue composition (muscle mass and fat mass). By measuring the body's muscle mass, fat mass and bone mineral density, one can estimate total body fat percentage.
Bone mineral density (BMD). | Measured 12 months postoperatively.
  Measured by DEXA scan.
KOOS | Measured 1 week before surgery.
  Knee - specific patient-reported outcome that measures the patient's own assessment of knee problems and related problems. The schedule consists of 42 questions representing 5 strands.
Pain | Measured 1 week before surgery.
  Visual Analogue Scale (VAS pain score)
Serum leptin. | Measured 1 week before surgery.
  Leptin is a hormone produced in fat tissue.
Heart rate | Measured 1 week before surgery.
  Cardiovascular complications.
Blood pressure | Measured 1 week before surgery.
  Cardiovascular complications.
6 minutes walk test (6MW). | Measured 8 week postoperatively.
  Used to target the operating level of the patient's daily activities.
6 minutes walk test (6MW). | Measured 12 months postoperatively
  Used to target the operating level of the patient's daily activities.
Body composition | Measured 8 week postoperatively
  Dual energy X-ray absorptiometry (DEXA) can measure total body bone mineral density and obtain accurate measurements of body tissue composition (muscle mass and fat mass). By measuring the body's muscle mass, fat mass and bone mineral density, one can estimate total body fat percentage.
Body composition | Measured 12 months postoperatively
  Dual energy X-ray absorptiometry (DEXA) can measure total body bone mineral density and obtain accurate measurements of body tissue composition (muscle mass and fat mass). By measuring the body's muscle mass, fat mass and bone mineral density, one can estimate total body fat percentage.
KOOS | Measured 8 week postoperatively
  Knee - specific patient-reported outcome that measures the patient's own assessment of knee problems and related problems. The schedule consists of 42 questions representing 5 strands.
KOOS | Measured 12 months postoperatively
  Knee - specific patient-reported outcome that measures the patient's own assessment of knee problems and related problems. The schedule consists of 42 questions representing 5 strands.
Pain | Measured 8 week postoperatively
  Visual Analogue Scale (VAS pain score)
Pain | Measured 12 months postoperatively
  Visual Analogue Scale (VAS pain score)
Serum leptin. | Measured 8 week postoperatively
  Leptin is a hormone produced in fat tissue.
Serum leptin. | Measured 12 months postoperatively
  Leptin is a hormone produced in fat tissue.
Heart rate | Measured 8 week postoperatively
  Cardiovascular complications.
Heart rate | Measured 12 months postoperatively
  Cardiovascular complications.
Blood pressure | Measured 8 week postoperatively
  Cardiovascular complications.
Blood pressure | Measured 12 months postoperatively
  Cardiovascular complications.

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, Prof. D.Msc, Principal Investigator — Department of Orthopedics Research Aarhus University Hospital
Locations (1):
- Department of Orthopedics Research Aarhus University Hospital, Aarhus, Denmark